CLINICAL TRIAL: NCT00081172
Title: A Phase II Trial Of Lu Radiolabeled Monoclonal Antibody HuJ591-GS (Lu-J591) In Patients With Metastatic Androgen-Independent Prostate Cancer
Brief Title: Radiolabeled Monoclonal Antibody in Treating Patients With Progressive Metastatic Androgen-Independent Adenocarcinoma (Cancer) of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: MSKCC-03144; CDR0000360629 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Radiation: lutetium Lu 177 monoclonal antibody J591

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver radioactive tumor-killing substances to them without harming normal cells.

PURPOSE: This phase II trial is studying how well radiolabeled monoclonal antibody works in treating patients with progressive metastatic androgen-independent adenocarcinoma (cancer) of the prostate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the prostate-specific antigen (PSA) response rate in patients with progressive metastatic androgen-independent adenocarcinoma of the prostate treated with lutetium Lu 177 monoclonal antibody J591.
* Determine the measurable disease response rate in patients treated with this drug.

Secondary

* Determine the toxicity of this drug in these patients.
* Determine the duration of biochemical PSA and/or measurable disease response in patients treated with this drug.
* Determine the incidence of human anti-J591 antibody (HAHA) response in patients treated with this drug.
* Correlate hematological toxicity of this drug with bone marrow involvement (bone scan index) in these patients.
* Determine the survival rate in patients treated with this drug.
* Determine the targeting of this drug to known tumor sites in these patients.
* Determine the tumor-absorbed radiation dose in patients treated with this drug.

OUTLINE: This is a multicenter, open-label study.

Patients receive a single dose of lutetium Lu 177 monoclonal antibody J591 IV on day 1. Patients then undergo radionuclide scanning between days 6-8 to confirm tumor targeting by the study drug.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 17-32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic disease
* Progressive disease after prior antiandrogen therapy, as evidenced by at least 1 of the following parameters:

  * New osseous lesions on bone scan
  * Greater than 25% increase in the sum of the products of the longest perpendicular diameters of the lesions OR the appearance of new lesions on MRI or CT scan
  * Rising prostate-specific antigen (PSA) despite adequate medical or surgical castration therapy

    * Consecutive increase in PSA, determined by two separate measurements taken at least 1 week apart and confirmed by a third, and if necessary, a fourth measurement
    * PSA must be ≥ 5 ng/mL and ≥ 25% above the previous nadir
* Measurable or evaluable disease
* Serum testosterone ≤ 50 ng/dL
* No confluent lesions involving axial and appendicular skeleton on bone scan ("superscan")

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Hematocrit ≥ 30%
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 150,000/mm^3
* No serious hematologic illness that would preclude study participation

Hepatic

* AST ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* PTT normal
* PT normal OR
* INR normal
* No serious hepatic illness that would preclude study participation

Renal

* Creatinine ≤ 2.5 mg/dL
* Calcium ≤ 11 mg/dL
* No serious renal illness that would preclude study participation

Cardiovascular

* No New York Heart Association class III or IV heart disease
* No active angina pectoris
* No prior deep vein thrombophlebitis within the past 3 months
* No other serious cardiac illness that would preclude study participation

Pulmonary

* No pulmonary embolus within the past 3 months
* No other serious respiratory illness that would preclude study participation

Other

* Fertile patients must use effective contraception
* HIV negative
* No serious CNS illness that would preclude study participation
* No active serious infection not controlled by antibiotics
* No other serious illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior red blood cell or platelet transfusions
* More than 2 weeks since prior hematopoietic growth factors
* No prior monoclonal antibody therapy except ProstaScint®
* No other concurrent monoclonal antibody-based therapy
* No concurrent medication to support platelet count (e.g., oprelvekin)

Chemotherapy

* More than 4 weeks since prior cytotoxic chemotherapy

Endocrine therapy

* See Disease Characteristics
* Concurrent luteinizing hormone-releasing hormone (LHRH) analog allowed provided 1 of the following is true:

  * Treatment is maintained during study participation
  * Treatment is terminated at least 10 weeks (for 1-month depot preparations), 24 weeks (for 3-month depot preparations), or 32 weeks (for 4-month depot preparations) prior to study entry
* More than 4 weeks since prior corticosteroids
* More than 4 weeks since prior adrenal hormone inhibitors
* Concurrent low-dose prednisone (≤ 5mg/day) for adrenal insufficiency allowed
* No concurrent finasteride

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25% of skeleton
* No prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium-containing compounds (e.g., Metastron® or Quadramet®)

Surgery

* Not specified

Other

* More than 4 weeks since prior PC-SPES
* More than 4 weeks since prior investigational therapy (medications or devices)
* At least 1 week since prior aspirin and/or nonsteroidal anti-inflammatory agents possessing antiplatelet activity
* At least 1 week since prior antiplatelet medication, including the following:

  * Abciximab
  * Cilostazol
  * Clopidogrel
  * Dipyridamole
  * Ticlopidine
* No concurrent anticoagulant medications (for platelet count < 50,000/mm^3), including the following:

  * Dalteparin
  * Danaparoid
  * Enoxaparin
  * Heparin
  * Warfarin
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Biochemical response as measured by prostate-specific antigen level at 8 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York